CLINICAL TRIAL: NCT05767333
Title: Evaluation of Cicaplast in Subjects With Skin Irritation for 21 Days
Brief Title: Evaluation of Cicaplast in Subjects With Skin Irritation
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: LRP21005-CICAPLAST BAUME B5
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Skin Diseases
Keywords: skin irritation; irritative dermatitis; superficial burn
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this open, before/after, multicentric study is to assess the effect and tolerance of Cicaplast Baume B5 in patients having a skin irritation (irritative and cracked dermatitis, dry eczematids, rubbing irritation, ...) under dermatological control. Patients are asked to apply the product at least twice a day until complete recovery (maximum 21 days).

DETAILED DESCRIPTION:
Dermscan has implemented a quality management system which has been certified by the International Standards Organization (ISO 9001: 2015). This quality assurance system includes appropriate Good Clinical Practices (GCP) and regulation requirements. The proofreader is not involved in the audited study. A certificate of quality inspection signed by the person who checked the report is enclosed in each study.

Statistical method

Regarding the descriptive analysis, the quantitative data is summarized using the following statistics by time point:

* Number of values
* Mean
* Median
* Standard deviation (SD)
* Minimum value
* Maximum value.

Are summarized in frequency (N) and percentage (%) by time point:

* the Investigator's Global Assessment (IGA) score assessed by the investigator using a 6-point scale
* the soothing effect assessed by the subject using a 4-point scale for the parameters pain and pruritus
* each global tolerance score assessed by the investigator and by the subject using a 4-point scale.

The score of anti-irritating effect (SCOre de REparation de l'EPIderme= SCOREPI) is summarized using statistics for quantitative variables at each time point.

The local signs of irritated area assessed using a 4-point scale (erythema, desquamation, pigmentation, cracks, oedema) are summarized in frequency (N) and percentage (%) and by time point and by parameter.

ELIGIBILITY:
Inclusion Criteria:

* subjects presenting the following skin irritations (at least 3 to 5 per irritation): irritative and cracked dermatitis, dry eczematids/dry patches, rubbing irritation in specific location (ex: thumb frictions, lichenifications), ...
* localization of irritation lesions: face, limbs, trunk, feet, fold, hands, ...
* subjects having a feeling of discomfort at the site of the lesion.

Exclusion Criteria:

* cutaneous pathology on the studied zone (other than the required irritations)
* use of topical or systemic treatment during the previous weeks liable to interfere with the assessment of the cutaneous acceptability of the study product (according to the investigator's appreciation);
* subject with healing disorder (keloid, hypertrophic)
* subject with Type 1 diabetic
* subject under chemotherapy and radiotherapy
* subject with a skin disease on evaluation site: psoriasis and atopic dermatitis active lesions and hand dermatitis

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: adults, teens and children meeting the inclusion and exclusion criteria and willing to adhere to the protocol and study procedures
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
evaluation of the effect on the recovery of irritated skin lesions | from baseline to Day21
  the investigator evaluates the improvement of the tested product using the IGA score on a 6-point scale (from -1: aggravation to 4: complete recovery)

SECONDARY OUTCOMES:
evaluation of the local signs of irritated area | from baseline to Day21
  the investigator assesses the local signs (erythema, desquamation, pigmentation, cracks, oedema) using a 4-point scale (from absent to severe)
evaluation of the anti-irritating effect | from baseline to Day21
  the investigator evaluates the lesions using SCOREPI tool which takes into account the following parameters: total surface of the skin lesions, erythema, desquamation, and cracks.
evaluation of the skin sensitivity | from baseline to Day21
  the patient evaluates the sensitivity of irritated areas using a 4-point scale for pain and pruritus ((from 0= absent to 3= severe)
evaluation of the global tolerance by the investigator | from baseline to Day21
  the investigator evaluates the global tolerance using a 4-point scale (from 0=null to 3= excellent)
evaluation of the global tolerance by the patient | from baseline to Day21
  the patient evaluates the global tolerance using a 4-point scale (from 0=null to 3= excellent)
evaluation of post-recovery marks | Day21
  the investigator assesses post-recovery marks score concerning type (redness, hyperpigmentation, hypopigmentation) and severity using a 4-point scale (from 1= almost absent to 4= severe) of an irritated area
evaluation of the global effect by the investigator | Day21
  the investigator evaluates the global effect using a 5-point scale (from -1= worsening to 3= excellent)
evaluation of the global effect by the patient | Day21
  the patient evaluates the global effect using a 5-point scale (from -1= worsening to 3= excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Le Floc'h, Study Director — Cosmetique Active International
Locations (4):
- EUROFINS CRL, Inc., Piscataway, New Jersey, United States
- EUROFINS CONSUMER PRODUCT TESTING Co. Ltd, Guangzhou, China
- Insight Research, Quatre Bornes, Mauritius
- EUROFINS DERMSCAN POLAND Sp., Gdansk, Poland